CLINICAL TRIAL: NCT05812053
Title: Comparative Evaluation of Eggshell Powder Versus Biodentine in Primary Teeth Pulpotomy: Clinical And Radiographic Study
Brief Title: Comparative Evaluation of Eggshell Powder in Primary Teeth Pulpotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #R-PED-9-20-2
Record Dates: First submitted 2023-03-21; First posted 2023-04-13 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pulpitis Reversible; Pulp Exposure, Dental
Keywords: Cone-beam computed tomography; egg shell powder; biodentine
MeSH Terms: conditions — Dental Pulp Exposure | interventions — Pulpotomy; Restraint, Physical

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1: Eggshell Powder (Experimental): 30 primary molars will be treated with Eggshell Powder freshly mixed with distilled water till it reaches a suitable consistency (1:1 ratio by volume) to cover pulp stumps
  Interventions: Procedure: pulpotomy; Radiation: cone beam computed tomography (CBCT) assessment
- group II: biodentine (Experimental): 30 primary molars will be treated with biodentine to cover pulp stumps
  Interventions: Procedure: pulpotomy; Radiation: cone beam computed tomography (CBCT) assessment
- group III: mineral tri-oxide aggregate (MTA) (Active Comparator): 30 primary molars will be treated with MTA to cover pulp stumps
  Interventions: Procedure: pulpotomy; Radiation: cone beam computed tomography (CBCT) assessment

INTERVENTIONS:
Procedure: pulpotomy — Teeth will be anesthetized then Rubber dam and high suction will be used in pulpotomy procedure. Cavity outline was performed by sterile #330 high speed bur using water spray. Caries was removed by large spoon excavator. When pulpal exposure occurred, the roof of pulp chamber removed by low speed round bur. Haemostasis was obtained by applying pressure with moist cotton pellet with saline. Then the test materials was applied. after that, pulp stumps of all molars in each group will be dressed using Intermediate restorative material then the tooth will be restored with a preformed stainless steel crown
Radiation: cone beam computed tomography (CBCT) assessment — a post-operative CBCT image will be taken immediately after completing the procedure with fixed exposure parameters (120 Kv, 5mA, and 0.125mm voxel size) using the smallest field of view (8D, 8Hcm) also, after 12 months follow-up periods.

SUMMARY:
To assess & compare clinical & radiographic effects of Eggshell Powder, Biodentine and MTA as pulpotomy agents in primary teeth.

DETAILED DESCRIPTION:
Pulpotomy is the most widely accepted technique for treating primary teeth with deep carious lesion, pulp exposure during the operatory process or after a traumatic pulp exposure. Mineral trioxide aggregate (MTA) is one such material that has shown tremendous potential for regeneration. Biodentine™ (hydraulic silicate cement) is a novel dental material with high mechanical characteristics as well as superior biocompatibility and bioactive behaviour. Nowadays, chicken eggshell powder (CESP) (a natural calcium-rich source) is achieving wide acceptance in the medical and dental fields. To date, there is insufficient evidence to properly evaluate Eggshell Powder as a pulpotomy agent in primary teeth; thus, the current study aimed to assess and compare clinical and radiographical success of Eggshell Powder, Biodentine and MTA as pulpotomy agents in primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* Restorable primary molars with deep carious lesions.
* Absence of gingival swelling or sinus tract.
* Absence of spontaneous pain
* Absence of pain on percussion.
* Absence of discontinuity of lamina dura
* Absence of internal root resorption.
* Absence of external root resorption.
* Absence of inter-radicular or periapical bone destruction (radiolucency).

Exclusion Criteria:

* presence of spontaneous pain
* presence of gingival swelling or sinus tract
* presence of internal or external root resorption
* pain on percussion.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
absence of pain | up to 12 months
  Measuring Method: Verbal Question to Patient /Parents Measuring Unite: score 0 for absence of pain and score 1 for presence of pain
absence of fistula | up to 12 months
  Measuring Method: Visual examination by operator Measuring Unite: score 0 for absence of swelling and score 1 for presence of swelling
Tenderness to percussion | Up to 12 month
  Measuring Method: Percussion test Measuring Unite: Binary (+/-)
Furcation radiolucency | 6 months
  Measuring Method: cone beam computed tomography (CBCT) for assessment of radio-density of bone at the furcation area Measuring Unite: Binary (+/-)
Furcation radiolucency | 12 months
  Measuring Method: cone beam computed tomography (CBCT) for assessment of radio-density of bone at the furcation area Measuring Unite: Binary (+/-)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Celik BN, Mutluay MS, Arikan V, Sari S. The evaluation of MTA and Biodentine as a pulpotomy materials for carious exposures in primary teeth. Clin Oral Investig. 2019 Feb;23(2):661-666. doi: 10.1007/s00784-018-2472-4. Epub 2018 May 10. PMID 29744721
- [Background] Nowicka A, Lipski M, Parafiniuk M, Sporniak-Tutak K, Lichota D, Kosierkiewicz A, Kaczmarek W, Buczkowska-Radlinska J. Response of human dental pulp capped with biodentine and mineral trioxide aggregate. J Endod. 2013 Jun;39(6):743-7. doi: 10.1016/j.joen.2013.01.005. Epub 2013 Apr 10. PMID 23683272
- [Background] Siva Rama Krishna D, Siddharthan A, Seshadri SK, Sampath Kumar TS. A novel route for synthesis of nanocrystalline hydroxyapatite from eggshell waste. J Mater Sci Mater Med. 2007 Sep;18(9):1735-43. doi: 10.1007/s10856-007-3069-7. Epub 2007 May 5. PMID 17483877
- [Background] Kattimani VS, Chakravarthi PS, Kanumuru NR, Subbarao VV, Sidharthan A, Kumar TS, Prasad LK. Eggshell derived hydroxyapatite as bone graft substitute in the healing of maxillary cystic bone defects: a preliminary report. J Int Oral Health. 2014 Jun;6(3):15-9. Epub 2014 Jun 26. PMID 25083027